CLINICAL TRIAL: NCT01481558
Title: Effects of Transcranial Direct Current Stimulation on the Apathy of Alzheimer's: a Randomized, Sham-controlled Clinical Trial
Brief Title: Effects of Transcranial Direct Current Stimulation on the Apathy of Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Claudia Kimie Suemoto, Assistant Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0679/11
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Results first posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Apathy; Alzheimer's Disease
Keywords: Apathy; Alzheimer's Disease; Dementia
MeSH Terms: conditions — Lethargy; Alzheimer Disease; Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham tDCS (Sham Comparator): sham-tDCS application every 2 days for 2 weeks (total of 6 applications)
  Interventions: Device: Transcranial direct current stimulation
- Transcranial direct current stimulation (Experimental): tDCS application every 2 days for 2 weeks (total of 6 applications)
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS 2 mA, dorsolateral pre-frontal cortex

SUMMARY:
This is a phase 2 double-blind, randomized, sham-controlled study to investigate the effects of repeated transcranial direct current stimulation for the treatment of apathy in moderate Alzheimer's Disease in patients selected from an outpatient clinics in São Paulo, Brazil.

DETAILED DESCRIPTION:
Forty patients were randomized to receive either active or sham-tDCS over the left dorsolateral prefrontal cortex (DLPFC). Patients received six sessions of intervention during two weeks and were evaluated at baseline, at week one and two, and after one week without intervention. Clinical raters, patients, and caregivers were blinded. The primary outcome was apathy. Global cognition and neuropsychiatric symptoms were examined as secondary outcomes.

ELIGIBILITY:
Inclusion criteria:

1. Dementia defined by DSM-IV (Diagnostic and Statistical Manual version IV)
2. Possible Alzheimer's Disease defined by NINCDS-ADRDA (National Institute for Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association)
3. Mini Mental State Examination scores from 10 to 20
4. Apathy defined by a score equal or higher to 14 in Apathy Scale

Exclusion criteria:

1. Clinical instability
2. Epilepsy
3. Metallic clip in the head
4. Use of alcohol and psychotropic drugs

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Study Director — Harvard Medical School (HMS and HSDM); Ricardo Nitrini, MD, PhD, Study Chair — University of Sao Paulo; Claudia K Suemoto, MD, PhD, Principal Investigator — University of Sao Paulo; Ester Nakamura-Palacios, MD, PhD, Study Chair — Federal University of Espirito Santo; Daniel Apolinário, MD, Study Chair — University of Sao Paulo
Locations (1):
- University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Suemoto CK, Apolinario D, Nakamura-Palacios EM, Lopes L, Leite RE, Sales MC, Nitrini R, Brucki SM, Morillo LS, Magaldi RM, Fregni F. Effects of a non-focal plasticity protocol on apathy in moderate Alzheimer's disease: a randomized, double-blind, sham-controlled trial. Brain Stimul. 2014 Mar-Apr;7(2):308-13. doi: 10.1016/j.brs.2013.10.003. Epub 2013 Oct 25. PMID 24262299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: January 2012 to May 2012 Location: Outpatient dementia clinic
Groups:
- Sham Transcranial Direct Current Stimulation: One application of sham tDCS every two days (total: 6 applications)
- Transcranial Direct Current Stimulation: One application of tDCS every two days (total: 6 applications)
Period: Overall Study
Arm/Group | Sham Transcranial Direct Current Stimulation | Transcranial Direct Current Stimulation
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Transcranial Direct Current Stimulation | Transcranial Direct Current Stimulation | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.6 (8.0) | 79.4 (7.1) | 80.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  Brazil | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Apathy Symptoms
Description: Apathy evaluated by Apathy Scale by Starsktein et al, 1992, which consists of 14 items phrased as questions that are to be answered by the caregiver on a four-point Likert scale. The total score range from 0 to 42, with higher scores indicating greater apathy severity. Apathy was assessed at baseline and at the end of the sixth session (second week).
Time Frame: Differences in outcome measure comparing second week to baseline
Population: alpha=5%, power=80%, SD estimated at 8 on Apathy scale scores, and correlation coefficient estimated at 0.7, a sample with 20 participants per arm is required to detect a between-group effect size of 0.5.
  Intention to treat (ITT) analyses were conducted using the method of last observation carried forward (LOCF) for missing data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sham Transcranial Direct Current Stimulation | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20 | 20
units on a scale | -2.05 [-3.68 to -0.42] | -1.95 [-3.49 to -0.41]
Statistical Analysis 1: Comparison: Sham Transcranial Direct Current Stimulation vs Transcranial Direct Current Stimulation; Test type: Superiority or Other; p = 0.55, ANCOVA; Mean Difference (Net) = 0.10, Standard Deviation 0.01

ADVERSE EVENTS:
Arm/Group | Sham Transcranial Direct Current Stimulation | Transcranial Direct Current Stimulation
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No